CLINICAL TRIAL: NCT04673331
Title: Comparison of Physical Activity, Exercise Capacity, Quality of Life, Cognitive Function and Coronavirus Phobia Levels of Adult Cystic Fibrosis Patients With Healthy Individuals With Telerehabilitation in the COVID-19 Pandemic
Brief Title: Physical Activity, Exercise Capacity and Coronavirus Phobia of Adult Cystic Fibrosis Patients During COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aydan Aslı Aksel Uylar, Physical Therapist, Hacettepe University
Other Study IDs: GO 20/794
Record Dates: First submitted 2020-12-12; First posted 2020-12-17 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic fibrosis: Inclusion Criteria:
  Having been diagnosed with cystic fibrosis Being over 18 years old The clinical condition is stable Having the ability to access the internet through a device (computer or mobile device) that enables video conferencing Giving consent on a voluntary basis
  Exclusion Criteria:
  Severe comorbidity that limits mobilization or physical activity(orthopedic, cardiac or neurological condition) Pregnancy
  Interventions: Other: exercise capacity
- Healthy individuals: Inclusion Criteria:
  Being over 18 years old Having the ability to access the internet through a device (computer or mobile device) that enables video conferencing Giving consent on a voluntary basis
  Exclusion Criteria:
  Severe comorbidity that limits mobilization or physical activity(orthopedic, cardiac or neurological condition) Pregnancy
  Interventions: Other: exercise capacity

INTERVENTIONS:
Other: exercise capacity — 3minute step test and 1minute sit to stand test used assessment of exercise capacity.

SUMMARY:
The purpose of this study was to evaluate physical activity, exercise capacity, quality of life, cognitive status level and coronavirus phobia level of adult cystic fibrosis patients and compare with the findings of healthy subjects with teleconference during COVID-19 pandemic.

DETAILED DESCRIPTION:
This study will be participated adult with cystic fibrosis and healthy individuals. Demographic information of individuals will be recorded in online video conference. Physical activity, exercise capacity and cognitive function levels will be measured during video conferencing.Then, the physical activity level, coronavirus phobia and quality of life of the participants will be evaluated subjectively with questionnaires through the Google forms.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old Having the ability to access the internet through a device (computer or mobile device) that enables video conferencing Giving consent on a voluntary basis

Exclusion Criteria:

* Severe comorbidity that limits mobilization or physical activity(orthopedic, cardiac or neurological condition) Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and healthy individuals between 18-65 years old, who are diagnosed with cystic fibrosis will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Physical Activity Level-International Physical Activity Questionnaire | 8 minutes
  Physical activity level will be evaluated International Physical Activity Questionnaire- Short Form (IPAQ-SF). IPAQ short version asks spended time during sitting, walking, moderate and vigorous physical activities. The score is obtained by multiplying the minutes, days and metabolic equivalent values. According to these scores, physical activity levels are classified as "inactive", "minimally active" and "very active".
Coronavirus Phobia-Coronavirus-19 Phobia Scale | 5 minutes
  COVID-19 phobia will be evaluated with Coronavirus-19 Phobia Scale (C19P-S) and total score ranges from 20-100. Lower scores mean better outcome.
Exercise Capacity | 15 minutes
  Exercise capacity will be evaluated with 1-minute sit to stand test and 3-minute step test. Maximum heart rate, minimum saturation, count of step are record during the 3 minute step test. Number of sit to stand for 1 minute is recorded end of the 1 minute sit to stand test.
Weekly Average Steps | 2 minutes
  The number of steps in the last week was recorded and averaged using the pedometer applications from the participants own smartphones.
  <5000 steps/day sedentary 5000-7499 steps/day low active 7500-9999 steps/day somewhat active
  ≥10 000 steps/day active >12 500 steps/day highly active

SECONDARY OUTCOMES:
Cognitive Function-Standardized Mini Mental State Examination | 5 minutes
  Cognitive function evaluation will be Standardized Mini Mental State Examination (SMMSE). Scores less than 23 mean cognitive impairment.
Quality Of Life-Nottingham Health Profile | 10 minutes
  Quality of life will be evaluated with Nottingham Health Profile (NHP). This questionnaire categorizes are energy, pain, emotional reactions, sleep, social isolation, physical mobility, depression and anxiety. Lower scores mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Naciye Vardar Yağlı, PhD, Study Director — Hacettepe University; Aydan Aslı Aksel, Principal Investigator — Hacettepe University; Ebru Damadoğlu, PhD, Study Chair — Hacettepe University; Merve Fırat, MSc, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided